CLINICAL TRIAL: NCT01802866
Title: A Phase 2b/3 Multicenter, Randomized, Double-Masked, Dose-Ranging Study Comparing the Efficacy and Safety of Emixustat Hydrochloride (ACU-4429) With Placebo for the Treatment of Geographic Atrophy Associated With Dry Age-Related Macular Degeneration
Brief Title: Safety and Efficacy Assessment Treatment Trials of Emixustat Hydrochloride
Acronym: SEATTLE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kubota Vision Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4429-202
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Geographic Atrophy
Keywords: Geographic atrophy; GA; Dry AMD
MeSH Terms: conditions — Geographic Atrophy | interventions — emixustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ACU-4429 2.5 mg (Experimental): 2.5 mg tablet
  Interventions: Drug: ACU-4429
- ACU-4429 5 mg (Experimental): 5 mg tablet
  Interventions: Drug: ACU-4429
- ACU-4429 10 mg (Experimental): 10 mg tablet
  Interventions: Drug: ACU-4429
- Placebo (Placebo Comparator): Includes identical tablets with only inactive ingredients (0 mg).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACU-4429 — Take orally once daily for 24 months
  Other Names: emixustat hydrochloride
  Arms: ACU-4429 10 mg; ACU-4429 2.5 mg; ACU-4429 5 mg
Drug: Placebo — Take orally once daily for 24 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if emixustat hydrochloride (ACU-4429) reduces the rate of progression of geographic atrophy compared to placebo in subjects with dry age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age ≥55 years.
2. Clinical diagnosis of GA associated with AMD
3. Able and willing to provide written informed consent.
4. Able to reliably administer oral medication by self or with available assistance.

Exclusion Criteria:

1. Active CNV or presence of an active ocular disease.
2. Known serious allergy to the fluorescein sodium for injection in angiography.
3. Pre-specified laboratory abnormalities at screening.
4. Treatment with any investigational study drug within 30 days of screening or device (within 60 days of screening)
5. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding
6. Female subjects who are pregnant or lactating.
7. Female subjects of childbearing potential and male subjects who are not surgically sterile who are not willing to practice a medically accepted method of birth control from screening through 30 days after completion of the study.
8. Unstable or poorly controlled medical or ophthalmic conditions

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2013-02; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the total area of the GA lesion(s) | 24 months

SECONDARY OUTCOMES:
Change from baseline in BCVA score | 24 months
Frequency of AEs, discontinuations due to AEs, or dose modifications; severity and seriousness of AEs | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Acucela Medical Monitor, Study Director — Kubota Vision Inc.
Locations (1):
- Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yeong JL, Loveman E, Colquitt JL, Royle P, Waugh N, Lois N. Visual cycle modulators versus placebo or observation for the prevention and treatment of geographic atrophy due to age-related macular degeneration. Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD013154. doi: 10.1002/14651858.CD013154.pub2. PMID 33331670
- [Derived] Rosenfeld PJ, Dugel PU, Holz FG, Heier JS, Pearlman JA, Novack RL, Csaky KG, Koester JM, Gregory JK, Kubota R. Emixustat Hydrochloride for Geographic Atrophy Secondary to Age-Related Macular Degeneration: A Randomized Clinical Trial. Ophthalmology. 2018 Oct;125(10):1556-1567. doi: 10.1016/j.ophtha.2018.03.059. Epub 2018 Apr 30. PMID 29716784